CLINICAL TRIAL: NCT07114042
Title: Moglobin, Albumin, Lymphocyte and Platelet Score as a Novel Predictor of Mortality and Re-bleeding in Patients With Upper Gastrointestinal Bleeding
Brief Title: HALP as a Novel Score for Prediction of Mortality and re_bleeding in Upper GIT Bleeding
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reham Refaat Baoumy, Resident doctor, Sohag University
Other Study IDs: Soh-med--25-7-11MS
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Upper endoscopy — Prediction of upper gastrointestinal r_bleeding and mortality

SUMMARY:
Evaluation of the prognostic utility of the HALP score in patients with upper gastrointestinal bleeding, particularly in predicting re_bleeding risk and mortality in internal medicine department in Sohag University Hospitals.

DETAILED DESCRIPTION:
Study for evaluation of the utility of hemoglobin, Albumin, Lymphocyte and Platelat score in prediction of mortality and re_bleeding in patient with upper gastrointestinal bleeding, Patients will be included if they were initially admitted to the emergency department, had a confirmed diagnosis of upper gastrointestinal bleeding via endoscopy, and were 18 years of age or older.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they were initially admitted to the emergency department, had a confirmed diagnosis of upper gastrointestinal bleeding via endoscopy, and were 18 years of age or older.

Exclusion Criteria:

* Incomplete clinical data.
* Lack of laboratory results obtained at emergency department admission necessary for the calculation of HALP score; albumin, hemoglobin (HGB), platelets (PLT), or international normalized ratio (INR).
* Pregnancy
* Patients with missing data on clinical outcomes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with upper gastrointestinal bleeding
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
"Mortality" | 6 months
Incidence of "Re_bleeding" | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Reham R Baeoumy, Master, Principal Investigator — Sohag
Locations (1):
- Faculty of Medicine -Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided